CLINICAL TRIAL: NCT04999345
Title: Effectiveness of Reconditioning Exercise on Mobility and Functional Recovery in Older Adults With Urinary Tract Cancer Following Curative Surgery
Brief Title: Effect of Reconditioning Exercise on Older Adults With Urinary Tract Cancer Following Curative Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng Kung University (Other)
Responsible Party: Principal Investigator, Pei-Yun Lee, Assistant professor, National Cheng Kung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A-ER-109-415
Record Dates: First submitted 2021-07-21; First posted 2021-08-10 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Rehabilitation
MeSH Terms: interventions — Rehabilitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Provide resistance and aerobic exercise
  Interventions: Other: Rehabilitation
- Control Group (Placebo Comparator): Health education and gross range of motion exercise for upper and lower extremities
  Interventions: Other: Health education

INTERVENTIONS:
Other: Rehabilitation — Progressive resistance exercise and graded aerobic exercise will be provided for those in the experimental group.
  Arms: Experimental Group
Other: Health education — Health education and gross joint range of motion exercise for bilateral upper and lower extremities will be provided for those in the control group.
  Arms: Control Group

SUMMARY:
As population ages, geriatric patients with urinary tract cancer suffer from more complications and functional decline that alter treatment plan despite advance in cancer surgery. It was found that these urinary tract cancer survivors required a longer time to recover to the state before the treatment, and some may be even unable to recover to the state before the treatment. Exercise intervention has been found to be beneficial to improve functional capacity for cancer survivors, such as breast cancer. However, it is unclear whether exercise intervention could also improve functional recovery and mobility in patients with urinary tract cancer following curative surgery, especially in older adults. The purpose of this study is to investigate the effect of reconditioning exercise on morbidity, oncological outcomes, and functional recovery in older adults with urinary tract cancer following curative surgery.

Patients aged over 65 years old and after having undergone curative surgery for confirmed urinary tract cancer will be recruited. The participants will be assigned into two groups using blocked randomization design. One group will receive reconditioning exercise training for five consecutive days, and the other group will receive exercise education. Structured questionnaire for comprehensive geriatric assessment and functional mobility, such as walking performance, will be used to assess the training effect. Outcome measures are assessed including major complication after surgeries, changes in functional status, tumor progression, and length of survival. Physical function measurement will include hand grip, muscle strength of lower extremities, and gait performance.

ELIGIBILITY:
Inclusion Criteria:

* after having undergone curative surgery for confirmed urinary tract cancer
* able to independently walk for at least 8 meters before surgery
* able to follow 3-step commands

Exclusion Criteria:

* having unstable medical conditions or metastasis
* having neuromuscular diseases, such as stroke, Parkinson's diseases
* unable to attend training sessions
* having other health issues which would interfere evaluation and exercise training

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2022-03-20 (Actual); Study Completion 2023-03-14 (Actual)

PRIMARY OUTCOMES:
Muscle strength of the lower extremities | Before training
  Muscle strength of bilateral hip flexor,knee extensor, ankle dorsiflexor, and ankle plantarflexor
Muscle strength of the lower extremities | After five-day training
  Muscle strength of bilateral hip flexor,knee extensor, ankle dorsiflexor, and ankle plantarflexor
Muscle strength of the lower extremities | Follow up at one month after training
  Muscle strength of bilateral hip flexor,knee extensor, ankle dorsiflexor, and ankle plantarflexor
Timed up and go test | Before training
  Subjects are asked to rise from a standard armchair, walk to a marker 3 m away, turn, walk back, and sit down again.
Timed up and go test | After five-day training
  Subjects are asked to rise from a standard armchair, walk to a marker 3 m away, turn, walk back, and sit down again.
Timed up and go test | Follow up at one month after training
  Subjects are asked to rise from a standard armchair, walk to a marker 3 m away, turn, walk back, and sit down again.
Six minute walk test | Before training
  Subjects are instructed to walk as far as possible for 6 minutes.
Six minute walk test | After five-day training
  Subjects are instructed to walk as far as possible for 6 minutes.
Six minute walk test | Follow up at one month after training
  Subjects are instructed to walk as far as possible for 6 minutes.

SECONDARY OUTCOMES:
Grip strength | Before training
  Hand grip strength will be measured with a handheld dynamometer.
Grip strength | After five-day training
  Hand grip strength will be measured with a handheld dynamometer.
Grip strength | Follow up at one month after training
  Hand grip strength will be measured with a handheld dynamometer.
Modified Katz Index of Independence in Activities of Daily Living | Before training
  Measure independence in basic activities of daily living, including bathing, dressing, toileting, transfers, continence, and feeding. Full score is 32. The lower the score indicates lower dependence in performing daily activities.
Modified Katz Index of Independence in Activities of Daily Living | After five-day training
  Measure independence in basic activities of daily living, including bathing, dressing, toileting, transfers, continence, and feeding. Full score is 32. The lower the score indicates lower dependence in performing daily activities.
Modified Katz Index of Independence in Activities of Daily Living | Follow up at one month after training
  Measure independence in basic activities of daily living, including bathing, dressing, toileting, transfers, continence, and feeding. Full score is 32. The lower the score indicates lower dependence in performing daily activities.
Lawton instrumental activities of daily living scale | Before training
  To assess more complex activities that allow an individual to live independently in a community, such as shopping, cooking, and managing finances. Full score is 24. The higher the score indicates better function in performing instrumental daily activities.
Lawton instrumental activities of daily living scale | After five-day training
  To assess more complex activities that allow an individual to live independently in a community, such as shopping, cooking, and managing finances. Full score is 24. The higher the score indicates better function in performing instrumental daily activities.
Lawton instrumental activities of daily living scale | Follow up at one month after training
  To assess more complex activities that allow an individual to live independently in a community, such as shopping, cooking, and managing finances. Full score is 24. The higher the score indicates better function in performing instrumental daily activities.
The Short Portable Mental Status Questionnaire (SPMSQ) | Before training
  To assess cognitive function, including tests of orientation, memory and recall the date, day of the week, place, telephone or address, birth date, current and etc.
The Short Portable Mental Status Questionnaire (SPMSQ) | After five-day training
  To assess cognitive function, including tests of orientation, memory and recall the date, day of the week, place, telephone or address, birth date, current and etc.
The Short Portable Mental Status Questionnaire (SPMSQ) | Follow up at one month after training
  To assess cognitive function, including tests of orientation, memory and recall the date, day of the week, place, telephone or address, birth date, current and etc.
The Short-form Geriatric Depression Scale (GDS) | Before training
  To measure depression. The scale consists of 15 questions with a full score of 15. Scores of 0-4 are considered normal; 5-8 indicate mild depression; 9-11 indicate moderate depression; and 12-15 indicate severe depression.
The Short-form Geriatric Depression Scale (GDS) | After five-day training
  To measure depression. The scale consists of 15 questions with a full score of 15. Scores of 0-4 are considered normal; 5-8 indicate mild depression; 9-11 indicate moderate depression; and 12-15 indicate severe depression.
The Short-form Geriatric Depression Scale (GDS) | Follow up at one month after training
  To measure depression. The scale consists of 15 questions with a full score of 15. Scores of 0-4 are considered normal; 5-8 indicate mild depression; 9-11 indicate moderate depression; and 12-15 indicate severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Yun Lee, PhD, Principal Investigator — National Cheng Kung University
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No